CLINICAL TRIAL: NCT02450409
Title: A New Technique to Produce Anatomical Alignment Results With Less Midflexion Instability in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Georg Matziolis, Prof. Dr. med., University of Jena
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REK_2015_1
Record Dates: First submitted 2015-05-11; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Total knee arthroplasty; Midflexion instability; Gap technique; Anatomical alignment
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- gap technique (GT) (Active Comparator): The patients receive a total knee arthroplasty using the established "gap technique" (gold standard serving as control). The intervention is the implantation of a total knee arthroplasty with this specific technique.
  Implantation of TKA using the gap technique is the intervention. Intervention is not a drug but a specific operative technique.
  Interventions: Procedure: Implantation of TKA using the gap technique
- anatomical alignment (AA) (Experimental): The patients receive a total knee arthroplasty using the new "anatomical alignment technique" (experimental). The intervention is the implantation of a total knee arthroplasty with this specific technique.
  Implantation of TKA using anatomical alignment Intervention is not a drug but a specific operative technique.
  Interventions: Procedure: Implantation of TKA using anatomical alignment

INTERVENTIONS:
Procedure: Implantation of TKA using the gap technique — Implantation of total knee arthroplasty using a specific operative technique (GT) serving as control.
  Arms: gap technique (GT)
Procedure: Implantation of TKA using anatomical alignment — Implantation of total knee arthroplasty using a specific operative technique (AA) being experimental.
  Arms: anatomical alignment (AA)

SUMMARY:
Beside the current standard of classical mechanical alignment of total knee replacements, increased interest is being shown in anatomical alignment. However, no surgical technique is capable of controlling the stability of the joint in midflexion. The purpose of the present study was to present and evaluate a new surgical technique, which aims to reduce the need for soft-tissue release and optimize stability in midflexion.

ELIGIBILITY:
Inclusion Criteria:

* The patients were to undergo surface replacement due to primary osteoarthritis of the knee

Exclusion Criteria:

* Joints that had undergone open surgery beforehand (e.g. high tibial osteotomy, fracture treatment) were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Measurement of midflexion instability (i.e. tibofemoral gap medially and laterally) in 30° and 60° of flexion | intraoperatively immediately before implantation of definite implants.
  The outcome measures are given in mm.

SECONDARY OUTCOMES:
performance of soft tissue release (yes / no) and extend of release if done. | intraoperatively
  The surgeon documents postoeperatively if a soft tissue release was done or not and what extend a release had.
  The outcome measure is given in numbers (0 ... 4).

OTHER OUTCOMES:
The Knee Society Score | 1 year postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich-Schiller University Jena, Campus Eisenberg, Eisenberg, Eisenberg, Germany